CLINICAL TRIAL: NCT00551174
Title: Open Label, Parallel Group, Multicenter Study of Two Intravenous (IV) Ibandronate Dose Regimens (2 mg Every 2 Months and 3 mg Every 3 Months) in Women With Postmenopausal Osteoporosis Who Completed Trial BM16550
Brief Title: A Study of Bonviva (Ibandronate) in Women With Post-Menopausal Osteoporosis Who Have Received Previous Bonviva Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA17904
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2011-05-30 (Estimated); Last update posted 2011-07-22 (Estimated); Status verified 2011-07

CONDITIONS: Post-Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Active Comparator)
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 3 mg IV every 3 months for 3 years. All patients received a minimum of calcium 500 milligrams/day (upper limit 1500 mg/day) and Vitamin D 400 Internation Units/day (IU/day).
  Arms: 1
Drug: ibandronate [Bonviva/Boniva] — 2 mg IV every 2 months for 3 years. All patients received a minimum of calcium 500 milligrams/day (upper limit 1500 mg/day) and Vitamin D 400 Internation Units/day (IU/day).
  Arms: 2

SUMMARY:
This 2-arm study was designed to assess the long-term safety and tolerability of intravenous (IV) treatment with 2 mg or 3 mg Bonviva in women with post-menopausal osteoporosis who had previously completed Bonviva study BM16550 (DIVA study; NCT00048074). Patients received Bonviva either 2 mg IV every 2 months, or 3 mg IV every 3 months. Patients also received daily supplementation with vitamin D and calcium. The anticipated time on study treatment was 2+ years, and the target sample size was 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of Bonviva study BM16550 (NCT00048074), with at least 75% compliance
* Ambulatory

Exclusion Criteria:

* Patients who completed the Bonviva study BM16550 (NCT00048074) >3 months before the planned start date for this study
* Malignant disease diagnosed since inclusion into previous study
* Treatment with drugs affecting bone metabolism since inclusion into previous study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2004-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (6):
  - Gainesville, Georgia
  - St Louis, Missouri
  - Omaha, Nebraska
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Madison, Wisconsin
- Australia (2):
  - St Leonards
  - Sydney
- Belgium (2):
  - Brussels
  - Liège
- Czechia (2):
  - Pilsen
  - Prague
- Denmark (5):
  - Aalborg
  - Aarhus
  - Ballerup Municipality
  - Copenhagen
  - Vejle
- France (2):
  - Lyon
  - Orléans
- Germany (3):
  - Berlin
  - Essen
  - Hamburg
- Budapest, Hungary
- Italy (3):
  - Arenzano
  - Siena
  - Valeggio sul Mincio
- Mexico (2):
  - Mexico City
  - Monterrey
- Norway (3):
  - Haugesund
  - Oslo
  - Stavanger
- Poland (2):
  - Grudziądz
  - Krakow
- South Africa (3):
  - Cape Town
  - Pretoria
  - Sommerset West
- Madrid, Spain
- Aberdeen, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrollment was to occur at centers that had participated in BM16550 (NCT00048074) in North America, Mexico, Europe, Australia, and South Africa.
Pre-assignment Details: Postmenopausal osteoporosis. Patients having completed study BM16550 (NCT00048074) and who had complied with the intravenous (IV) regimen during the second year of study BM16550 (NCT00048074) for 75% or more.
Groups:
- 2 mg Ibandronate q2mo: 2 mg ibandronate intravenously (IV) every 2 months (q2mo) for 3 years
- 3 mg Ibandronate q3mo: 3 mg ibandronate intravenously (IV) every 3 months (q3mo) for 3 years
Period: Overall Study
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo
Started | 381 | 400
Completed | 362 (Intent-to-Treat (ITT) Population) | 394 (Intent-to-Treat (ITT) Population)
Not Completed | 19 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo | Total
Number analyzed (Participants) | 381 | 400 | 781
Age Continuous [Mean (Standard Deviation); unit: years] | 68.2 (6.1) | 67.9 (6.0) | 68.0 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 381 | 400 | 781
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 363 | 388 | 751
  Black | 0 | 0 | 0
  Oriental | 0 | 0 | 0
  Hispanic | 17 | 11 | 28
  Other | 1 | 1 | 2
BMI [Mean (Standard Deviation); unit: kg/m*2] | 25.63 (4.295) | 25.89 (4.394) | 25.76 (4.3460)

OUTCOME MEASURES:

1. Primary Outcome: Relative Percent Change From Baseline in Mean Lumbar Spine Bone Mineral Density (BMD) at 12, 24 and 36 Months
Description: Relative change percent(%) from baseline of MA17904 and BM16550 (NCT00048074) in mean lumbar spine (L2-L4) BMD at 12, 24 and 36 months (i.e., 3, 4 and 5 years after initiation of BM16550)- Study MA17940.Percent change=[(measure at time t - measure at baseline)/measure at baseline]*100%, where t=12, 24 and 36 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline,12, 24 and 36 months
Population: ITT population: 3 mg group = 394, 2 mg group = 362. Analysis populations (AP) for Month 12: 3 mg group = 383, 2 mg group = 348; Month 24: 3 mg group = 374, 2 mg group = 332; Month 36: 3 mg group = 349, 2 mg group = 314.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo
Number analyzed (Participants) | 362 | 394
Percent change
  Baseline | 0.7969 (0.0764) | 0.7861 (0.0824)
  Percent Change from Baseline at Month 12 | 0.8378 (3.1920) | 0.8845 (3.6386)
  Percent Change from Baseline at Month 24 | 1.6785 (3.6494) | 1.5742 (4.0665)
  Percent Change from Baseline at Month 36 | 1.9813 (4.6619) | 2.0559 (4.4747)

2. Secondary Outcome: Relative Percent Change From Baseline in Mean Total Hip BMD at 12, 24 and 36 Months
Description: Relative change percent (%) from baseline of MA17904 and BM16550 (NCT00048074) in mean total hip BMD at 12, 24 and 36 months (i.e., 3, 4 and 5 years after initiation of BM16550)- Study MA17904. Percent change=[(measure at time t - measure at baseline)/measure at baseline]*100%, where t=12, 24 and 36 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline,12, 24 and 36 months
Population: ITT populations: 3 mg group = 394, 2 mg group = 362. Analysis populations (AP) for Month 12: 3 mg group = 381, 2 mg group = 347; Month 24: 3 mg group = 371, 2 mg group = 330; Month 36: 3 mg group = 349, 2 mg group = 314.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo
Number analyzed (Participants) | 362 | 394
Percent change
  Baseline | 0.7651 (0.1035) | 0.7665 (0.0954)
  Percent Change from Baseline at Month 12 | 0.4487 (2.5604) | 0.1258 (3.0450)
  Percent Change from Baseline Month 24 | 0.0483 (3.0148) | -0.049 (3.0440)
  Percent Change from Baseline at Month 36 | -0.1546 (3.3604) | -0.2619 (4.0099)

3. Secondary Outcome: Relative Percent Change From Baseline in Serum C-telopeptide Crosslinks of Type I Collagen (CTX) at Trough at 6, 12, 24 and 36 Months
Description: Relative percent (%) change from baseline of MA17904 and BM16550 (NCT00048074) in serum C-telopeptide crosslinks of type I collagen (CTX) at trough at 6, 12, 24 and 36 months- Study MA17904. Percent change=[(measure at time t - measure at baseline)/measure at baseline]*100%, where t=6, 12, 24 and 36 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline, 6, 12, 24 and 36 months (i.e., 2.5, 3, 4 and 5 years after initiation of BM16550)
Population: Per-Protocol population: 3 mg group = 363, 2 mg group = 344. Analysis populations (AP) for Month 6: 3 mg group = 87, 2 mg group: 92; Month 12: 3 mg group = 92, 2 mg group = 92; Month 24: 3 mg group = 83, 2 mg group = 85; Month 36: 3 mg group = 75, 2 mg group = 76.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo
Number analyzed (Participants) | 344 | 363
Percent change
  Baseline | 0.232 (0.1327) | 0.264 (0.1497)
  Percent Change from Baseline at Month 6 | 17.562 (64.2113) | 20.091 (65.6960)
  Percent Change from Baseline at Month 12 | 35.934 (82.8825) | 34.009 (103.5972)
  Percent Change from Baseline at Month 24 | 42.237 (73.7395) | 47.442 (121.5415)
  Percent Change from Baseline at Month 36 | 41.478 (67.1965) | 58.478 (160.1702)

4. Secondary Outcome: Relative Percent Change From Baseline in Post-dose Suppression of Serum CTX at 6 Months
Description: Relative percent (%) change from MA17904 baseline of post-dose suppression of serum C-telopeptide crosslinks of type I collagen (CTX) at 6 months- Study MA17904. Percent change=[(measure at time t - measure at baseline)/measure at baseline]*100%, where t= 6 months. The baseline value is used as a reference to calculate the relative change from baseline.
Time Frame: Baseline, 6 months
Population: Per-Protocol population: 3 mg group = 363, 2 mg group = 344. Analysis populations (AP) for Month 6: 3 mg group = 89, 2 mg group: 93.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo
Number analyzed (Participants) | 344 | 363
Percent change
  Baseline | 0.232 (0.1327) | 0.264 (0.1497)
  Percent Change from Baseline at Month 6 | -78.024 (18.2619) | -81.617 (22.0440)

ADVERSE EVENTS:
Arm/Group | 2 mg Ibandronate q2mo | 3 mg Ibandronate q3mo
Serious Adverse Events (participants affected / at risk) | 90/381 | 84/400
Other Adverse Events (participants affected / at risk) | 265/381 | 285/400
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg Ibandronate q2mo (N=381) | 3 mg Ibandronate q3mo (N=400)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 5
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Radius Fracture (Injury, poisoning and procedural complications) | 3 | 2
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 3
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 2
Ulna Fracture (Injury, poisoning and procedural complications) | 1 | 2
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 | 0
Pneumonia (Infections and infestations) | 5 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Foot Deformity (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2
Myocardial Infarction (Cardiac disorders) | 6 | 0
Atrial Fibrillation (Cardiac disorders) | 3 | 0
Myocardial Ischaemia (Cardiac disorders) | 2 | 1
Hiatus Hernia (Gastrointestinal disorders) | 1 | 2
Transient Ischaemic Attack (Nervous system disorders) | 1 | 3
Cerebrovascular Accident (Nervous system disorders) | 0 | 3
Sciatica (Nervous system disorders) | 2 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Uterine Polyp (Reproductive system and breast disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Vertigo (Ear and labyrinth disorders) | 3 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma Pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign Uterine Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous Cell Carcinoma of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 1 | 1
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hand Fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon Rupture (Injury, poisoning and procedural complications) | 1 | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Borrelia Infection (Infections and infestations) | 1 | 0
Breast Abscess (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Escherichia Bacteraemia (Infections and infestations) | 0 | 1
Eye Infection (Infections and infestations) | 0 | 1
Gallbladder Empyema (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Herpes Zoster Ophthalmic (Infections and infestations) | 0 | 1
Infective Tenosynovitis (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 1 | 0
Typhoid Fever (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Flutter (Cardiac disorders) | 0 | 1
Atrioventricular Block Complete (Cardiac disorders) | 0 | 1
Cardiac Discomfort (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 1
Coronary Artery Disease (Cardiac disorders) | 1 | 0
Left Ventricular Failure (Cardiac disorders) | 1 | 0
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 1 | 0
Duodenal Ulcer (Gastrointestinal disorders) | 1 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Femoral Hernia (Gastrointestinal disorders) | 0 | 1
Gatritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal Disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 | 0
Pancreatitis Necrotising (Gastrointestinal disorders) | 1 | 0
Papilla of Vater Stenosis (Gastrointestinal disorders) | 1 | 0
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Carotid Artery Stenosis (Nervous system disorders) | 1 | 0
Cauda Equina Syndrome (Nervous system disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
Parkinson's Disease (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vaginal Haemorrhage (Reproductive system and breast disorders) | 1 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 1 | 0
Uterine Prolapse (Reproductive system and breast disorders) | 1 | 0
Vaginal Prolapse (Reproductive system and breast disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Malaise (General disorders) | 0 | 1
Multi-Organ Failure (General disorders) | 1 | 0
Non-Cardiac Chest Pain (General disorders) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Bile Duct Stone (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Urethral Stenosis (Renal and urinary disorders) | 1 | 0
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1
Dacryostenosis Acquired (Eye disorders) | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Platelet Count Decreased (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 mg Ibandronate q2mo (N=381) | 3 mg Ibandronate q3mo (N=400)
Nasopharyngitis (Infections and infestations) | 79 | 67
Back Pain (Musculoskeletal and connective tissue disorders) | 64 | 71
Hypertension (Vascular disorders) | 53 | 59
Arthralgia (Musculoskeletal and connective tissue disorders) | 57 | 47
Influenza (Infections and infestations) | 42 | 44
Hypercholesterolaemia (Metabolism and nutrition disorders) | 36 | 31
Bronchitis (Infections and infestations) | 33 | 27
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 29 | 27
Urinary Tract Infection (Infections and infestations) | 31 | 23
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 31 | 21
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 25 | 27
Pneumonia (Infections and infestations) | 21 | 24
Cystitis (Infections and infestations) | 24 | 18
Diarrhoea (Gastrointestinal disorders) | 21 | 21
Cataract (Eye disorders) | 19 | 21
Upper Respiratory Tract Infection (Infections and infestations) | 20 | 20
Depression (Psychiatric disorders) | 15 | 21
Dizziness (Nervous system disorders) | 21 | 8
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 20 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.